CLINICAL TRIAL: NCT05416320
Title: A Pilot Study of Calcipotriol as a Novel Treatment for Central Centrifugal Cicatricial Alopecia
Brief Title: Calcipotriol as a Novel Treatment for Central Centrifugal Cicatricial Alopecia (CCCA)
Acronym: CCCA
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The IRB was closed without enrolling any participants
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076702
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Central Centrifugal Cicatricial Alopecia
Keywords: hair loss; hair follicle regrowth
MeSH Terms: conditions — Alopecia | interventions — calcipotriene

STUDY DESIGN:
Intervention Model Description: 10 patients for the study will be randomized to one of two groups who consent to participate in a novel treatment with calcipotriol, or the control (no additional treatment besides Subject's already prescribed drug)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcipotriol Group (Experimental): Subjects will use the topical formulation once daily on the scalp. The subjects will use the treatment for a total of 6 months.
  Interventions: Drug: Calcipotriol
- Control Group (Sham Comparator): Subjects will continue to use their primary physician prescribed topical formulation once daily on the scalp. The subjects will use their treatment for a total of 6 months.
  Interventions: Drug: Subject's already prescribed drug

INTERVENTIONS:
Drug: Calcipotriol — Subjects will use the topical formulation once daily on the scalp. The subjects will use the treatment for a total of 6 months.
  Other Names: Dovonex
  Arms: Calcipotriol Group
Drug: Subject's already prescribed drug — Subjects will continue to use their already prescribed topical formulation once daily on the scalp. The subjects will use their treatment for a total of 6 months.
  Arms: Control Group

SUMMARY:
The purpose of this pilot study is to determine if calcipotriol shows potential to be an effective treatment for Central Centrifugal Cicatricial Alopecia (CCCA). This study aims to evaluate calcipotriol due to the possible anti-inflammatory effects that may affect the hair growth cycle.

DETAILED DESCRIPTION:
Calcipotriol, a vitamin D analog, has been topically used to treat alopecia areata, a form of non-scarring autoimmune alopecia in several studies. It is possible that Vitamin D plays a role in sustaining the hair follicle's immune privilege through anti-inflammatory effects such as controlling Interferon gamma (IFN-γ) production. A recent study showed a significant decrease of vitamin D in Black patients with Central Centrifugal Cicatricial Alopecia (CCCA)"

ELIGIBILITY:
Inclusion Criteria:

* Women who are eighteen years of age or older
* biopsy-proven and/or clinical diagnosis of CCCA Stage II-IV
* must be on stable treatment without changes for at least 3 months
* Subjects will be recruited from outpatient dermatology clinics at the Wake Forest Baptist Health Department of Dermatology.

Exclusion Criteria:

* Males

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males are excluded from this study since the prevalence of CCCA in males is so significantly low that it is difficult to find cases in a clinical setting
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Amount of hairline stabilization | Baseline
  Standardized camera and dermatoscopic photographs
Amount of hairline stabilization | Month 2
  Standardized camera and dermatoscopic photographs
Amount of hairline stabilization | Month 4
  Standardized camera and dermatoscopic photographs
Amount of hairline stabilization | Month 6
  Standardized camera and dermatoscopic photographs

SECONDARY OUTCOMES:
Amount of hair regrowth | Baseline, Month 2, Month 4, and Month 6
  Standardized camera and dermatoscopic photographs
Signs and symptoms of disease score | Month 2, Month 4, and Month 6
  standardized questionnaire - higher scores denotes worse condition
Dermatology Life Quality Index score | Baseline and Month 6
  scores of "not at all" to "very much"

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No